CLINICAL TRIAL: NCT06084364
Title: Painful Inflammatory Carpometacarpal-1 Osteoarthritis Treated With Intraarticular Steroids, Saline or an Occupational Therapy Intervention: the PICASSO Trial.
Brief Title: Intraarticular Steroids, Saline and Occupational Therapy in People With CMC1 Osteoarthritis
Acronym: PICASSO
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Collaborators: Vestre Viken Hospital Trust (Other); Helse Stavanger HF (Other Government); Haugesund Rheumatism Hospital (Other); St. Olavs Hospital (Other); Nordlandssykehuset HF (Other)
Responsible Party: Principal Investigator, Ida Kristin Haugen, Rheumatologist, senior researcher, Diakonhjemmet Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-505254-17-00
Record Dates: First submitted 2023-10-11; First posted 2023-10-16 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Osteoarthritis Thumb
Keywords: thumb; pain; inflammation; steroids; RCT; Occupational Therapy; Carpometacarpal-1; HappyHands; CMC-1; Picasso; intraarticular corticosteroid injections; IACS injections; thumb base pain; triamcinolone acetonide; Kenacort-T; osteoarthritis; OA
MeSH Terms: conditions — Pain; Inflammation; Osteoarthritis | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participants and the occupational therapist who examine the patients are blinded for the content of the intraarticular injections. The rheumatologist who perform the intraarticular injection will not be blinded for the content.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intraarticular corticosteroid injection (IACS) (Experimental): A single ultrasound-guided intraarticular injection of 0.50 ml of 40 mg/ml triamcinolone acetonide at baseline. A smaller dosage can be considered if there is increased resistance during injection. The same injection procedure will be repeated after 12 weeks if there is pain (NRS≥3) and inflammation (grey scale synovitis grade 1-3) present in the CMC-1 joint.
  Interventions: Drug: Injection of triamcinolone acetonide into the CMC-1 joint
- Saline injection (Placebo Comparator): A single ultrasound-guided intraarticular injection of 0.50 ml of sodium chloride 9 mg/ml at baseline. A smaller dosage can be considered if there is increased resistance during injection. The same injection procedure will be repeated after 12 weeks if there is pain (NRS≥3) and inflammation (grey scale synovitis grade 1-3) present in the CMC-1 joint.
  Interventions: Drug: Placebo
- Occupational Therapy intervention (Experimental): Patient education, instructions about hand exercises and training in the Happy Hands app. Administration of day and night orthosis. The Happy Hands app involves a 12 week intervention.
  Interventions: Behavioral: Multimodal Occupational therapy for CMC-1 joint OA

INTERVENTIONS:
Drug: Injection of triamcinolone acetonide into the CMC-1 joint — intraarticular injection with triamcinolone acetonide
  Other Names: Kenacort-T 40 mg/ml
  Arms: Intraarticular corticosteroid injection (IACS)
Behavioral: Multimodal Occupational therapy for CMC-1 joint OA — Patient education, instructions about hand exercises, orthosis and training
  Arms: Occupational Therapy intervention
Drug: Placebo — Intraarticular injection with saline
  Other Names: Sodium chloride 9 mg/ml
  Arms: Saline injection

SUMMARY:
A placebo-controlled randomized controlled trial exploring the effect of intraarticular steroids, saline or an occupational therapy intervention in inflammatory carpometacarpal-1 osteoarthritis

DETAILED DESCRIPTION:
The primary aim of the PICASSO trial is to examine the efficacy and safety of intraarticular corticosteroid injections and a multimodal occupational therapy intervention in patients with CMC-1 OA (Phase 1). By comparing available non-pharmacological and pharmacological treatments head-to-head, our results will be of interest to the range of health professionals who are involved in the management of CMC-1 OA patients. By including patients who are likely to benefit from the intervention (painful and inflammatory CMC-1 OA), appropriate dosage of drug and ultrasound-guided injections, our trial is more guarded against possible false negative results than previous studies. We will also explore predictors for treatment effects. Due to the heterogeneous presentation of OA, it is unlikely that one treatment will fit all, and treatment should be tailored to the patients´ clinical presentation. Second, we will explore the long-term safety of IACS, and whether the occupational therapy intervention can prevent or halt CMC-1 subluxation (Phase 2).

ELIGIBILITY:
Inclusion Criteria:

- Adult (40-85 years of age) men and women

In target CMC-1 joint:

* OA confirmed by radiographs or ultrasound examination, and
* Inflammation by ultrasound (grey scale synovitis grade 1-3), and
* Pain of at least 3 on a 0-10 Numeric Rating Scale (NRS) at rest or during activities at both pre-screening and screening.
* Patient is assessed as eligible for the proposed use of Kenacort-T

Exclusion Criteria:

* Use of thumb orthosis on most of the days or structured hand exercises in the last 12 weeks
* Intraarticular injections in the target CMC-1 joint in the last 12 weeks
* More than 3 previous IACS in the target CMC-1 joint
* Use of oral, intramuscular or intravenous steroids in the last 12 weeks
* Previous surgery of the target CMC-1 joint
* Planned hand surgery in the coming 24 weeks
* Do not want to quit using oral or topical NSAIDs on the hands (such as ibuprofen, diclofenac, etoricoxib, naproxen) in the next 12 weeks
* Systemic inflammatory joint diseases (such as rheumatoid arthritis (RA), psoriatic arthritis or gout) or other conditions that can better explain the hand pain (such as thoracic outlet syndrome, carpal tunnel disease, diabetic cheiropathy, hand injury in previous six months, or palmar tenosynovitis/trigger finger)
* Diagnosis of fibromyalgia
* Diagnosis of psoriasis
* Infection, skin disease or wounds at joint injection site
* Serious comorbidities, cognitive dysfunction, substance/alcohol abuse or any other medical condition that makes adherence to the study protocol difficult
* Severe or uncontrolled infections
* Known hypersensitivity to Triamcinolone acetonide (Kenacort) or any of the excipients (sodium carboxymethylcellulose, sodium chloride, polysorbate, benzyl alcohol, sodium hydroxide or hydrochloric acid)
* Included in another clinical study
* Use of digitalis glycosides
* Patients vaccinated or immunized with live virus vaccines in the last 2 weeks
* Not being able to talk or understand Norwegian
* Known pregnancy or planned pregnancy in the next 6 months
* Any condition that in the view of the investigator would suggest that the patient is unable to comply with the study protocol and procedures

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Estimated)
Dates: Start 2023-11-03 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Pain during activities in thumb base joint | 4 and 12 weeks
  Change in thumb base joint pain during activities last 24 hours on a 0-10 Numeric Rating Scale (NRS). 0 being no pain and 10 being the worst pain imaginable.

SECONDARY OUTCOMES:
Pain during activities in thumb base joint | All visits
  Change in thumb base joint pain during activities last 24 hours on a 0-10 Numeric Rating Scale (NRS). 0 being no pain and 10 being the worst pain imaginable.
Pain at rest in thumb base joint | Week 00, 04, 12, 24, 104
  Change in thumb base joint pain at rest last 24 hours on a 0-10 Numeric Rating Scale (NRS). 0 being no pain and 10 being the worst pain imaginable.
Pain during activities in finger joints | Week 00, 04, 12, 24, 104
  Change in finger joint pain during activities last 24 hours on a 0-10 Numeric Rating Scale (NRS). 0 being no pain and 10 being the worst pain imaginable.
Pain at rest in finger joints | Week 00, 04, 12, 24, 104
  Change in finger joint pain in rest last 24 hours on a 0-10 Numeric Rating Scale (NRS). 0 being no pain and 10 being the worst pain imaginable.
AUSCAN (Australian/Canadian hand index) | Week 00, 04,12, 24 and 104
  Change in Australian/Canadian Osteoarthritis Hand Index (AUSCAN) pain, stiffness and function subscales. Sum scores for pain (range: 0-20), stiffness (range: 0-4) and function (range: 0-36) can be calculated with higher scores representing worse health.
OMERACT-OARSI criteria responders | Week 00, 04, 12, 24, 104
  Number of OMERACT-OARSI criteria responders
MAP-Hand | Week 00, 04,12, 24 and 104
  Change in measure of activity performance of the hand
Patient-reported overall disease activity | Week 00, 04, 12, 24, 104
  Change in patient-reported overall disease activity in hands last 24 hours on a 0-10 Numeric Rating Scale (NRS). 0 being no disease activity and 10 being the worst disease activity imaginable.
Assessor-reported overall disease activity | Week 00, 04, 12, 24, 104
  Change in assessor-reported overall disease activity in hands on a 0-10 Numeric Rating Scale (NRS). 0 being no disease activity and 10 being the worst disease activity imaginable.
Pain in finger joints (hand figure) | Week 00, 04, 12, 24, 104
  Change in pain in finger joints last 24 hours (hand figure)
Grip strength | Week 00, 04, 12, 24, 104
  Change in grip strength
Use of analgesics | Week 00, 04, 12, 24, and 104
  Change in use of analgesics
Use of NSAIDs | Week 00, 04, 12, 24, and 104
  Change in use of non-steroidal anti-inflammatory drugs (NSAIDs)
Arthritis self-efficacy scale | Week 00, 04, 12, 24, 104
  Change in arthritis self-efficacy scale. The response categories are 10-100 with 10 points increment between each response category. A sum score is created based on the average of the five questions. Higher scores represent better self-efficacy.
Patient satisfaction | Week 04, 12
  Number of responders regarding self-reported perceived effect of treatment (yes/no). Patient satisfaction will be assessed with a question about whether the participants believe that they have had effect of the received treatment.
EuroQol 5 dimensions 5-levels (EQ-5D-5L) | Week 00, 04, 12, 24,104
  Change in EuroQol 5 dimensions 5-levels (EQ-5D-5L). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. On the EQ-VAS the participant is instructed to self-rate their health on a 0-100 scale, where 0=worst health and 100=best health.
Tender hand joints | Week 00, 04, 12, 24, 104
  Change in number of tender hand joints
Swollen hand joints | Week 00, 04, 12, 24, 104
  Change in number of swollen hand joints
Ultrasound synovitis in the CMC-1 joint | Week 00, 04,12, 24, 104. Will also be assessed in relation to additional injections in Phase 2.
  Change in ultrasound synovitis in the CMC-1 joint
Synovitis in the CMC-1 joint | Week 00, 04
  Change in MRI synovitis in the CMC-1 joint on contrast-enhanced MRI
Bone marrow lesions in the CMC-1 joint | Week 00, 04
  Change in bone marrow lesions in the CMC-1 joint on contrast-enhanced MRI
Structural progression | Week 00, 104
  Change in structural progression by Kellgren-Lawrence
Osteophytes | Week 00, 104
  Change in osteophytes by OARSI atlas
Joint space narrowing | Week 00, 104
  Change in joint space narrowing by OARSI atlas
Subluxation of the CMC-1 joint | Week 00, 104
  Change in subluxation of the CMC-1 joint
Adverse events | Week 00, 04, 12, 24, 104. Will also be assessed in relation to additional injections in Phase 2.
  Number of adverse events
Serious adverse events | Week 00, 04, 12, 24, 104. Will also be assessed in relation to additional injections in Phase 2.
  Number of serious adverse events
Withdrawals because of adverse events | Week 04, 12, 24, 104. Will also be assessed in relation to additional injections in Phase 2.
  Number of withdrawals because of adverse events
Use of healthcare services | Week 00, 12, 24, 104
  Questions about use of healthcare services

CONTACTS AND LOCATIONS:
Overall Officials: Ida Kristin Haugen, MD, PhD, Study Director — Diakonhjemmet Hospital; Marte Ingeborg Sæther, Principal Investigator — Martina Hansens Hospital; Elisabet Esperø, Principal Investigator — Haugesund Rheumatism Hospital; Katrine Brække Norheim, Principal Investigator — Helse Stavanger HF; Mari Hoff, Principal Investigator — St. Olavs Hospital; Göran Karlsson, Principal Investigator — Nordland Hospital
Locations (6):
- Norway (6):
  - Nordlands Hospital, Bodø
  - Haugesund Rheumatism Hospital, Haugesund
  - Diakonhjemmet Hospital, Oslo
  - Martina Hansens Hospital, Sandvika
  - Stavanger University Hospital, Stavanger
  - St Olavs Hospital, Trondheim

REFERENCES:
- [Derived] Gloersen M, Kjeken I, Tveter AT, Kazemi A, Sexton J, Dziedzic K, Felson DT, Stamm TA, Guermazi A, Hermann-Eriksen M, Saether MI, Lundby K, Espero EL, Olsen M, Norheim KB, Fister EB, Hoff M, Uleberg JK, Midtgard IP, Andreassen T, Sjolie D, Sletten H, Hammer HB, Haugen IK; PICASSO study team. Study protocol for the PICASSO trial: A randomized placebo-controlled trial to investigate the efficacy and safety of intraarticular steroid injections and an occupational therapy intervention in painful inflammatory carpometacarpal-1 osteoarthritis. Osteoarthr Cartil Open. 2024 Nov 19;7(1):100542. doi: 10.1016/j.ocarto.2024.100542. eCollection 2025 Mar. PMID 39669005